CLINICAL TRIAL: NCT06922266
Title: Personalizing Adoptive Cell Transfer for Solid Tumors: Towards a New Patient-tailored Treatment Option
Acronym: Chewbacca
Status: Not yet recruiting | Type: Observational
Sponsor: Ospedale San Raffaele (Other)
Collaborators: Fondazione Umberto Veronesi (Other)
Responsible Party: Principal Investigator, Chiara Maria Cattaneo, PhD, Ospedale San Raffaele
Other Study IDs: Chewbacca
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Immunotherapy; Precision Oncology; Lung cancer; Adoptive Cell Transfer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Tissue and blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Non-small cell lung cancer (NSCLC) patients: Adult subjects with diagnosis of non-small cell lung cancer (NSLC) that could undergo surgery or neo-adjuvant treatment.

SUMMARY:
This is a monocentric prospective observational study. This study will include patients with a diagnosis of non-small cell lung cancer for the collection of blood and tissue specimens.

DETAILED DESCRIPTION:
This study seeks to advance patient-specific cancer immunotherapy, through the ex-vivo generation of tumor-specific T cells recognizing and targeting tumor-specific mutations.

The study will enroll 20 adult patients with a diagnosis of non-small cell lung cancer, including those with lymph node involvement. Biological samples, including tumor and healthy lung tissue, as well as peripheral blood, will be collected pre-surgery and pre-treatment. The establishment of this sample collection will enable the detailed study of tumor-specific immune responses in non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to provide informed consent for participation in the study.
* Age: Adults aged 18 years or older.
* Diagnosis: non-small cell lung cancer (Stage I-II, III), with or without lymph node involvement, ideally with sufficient tumor burden to provide adequate tissue for analysis. In accordance with good clinical practice, patients with early-stage disease will undergo direct surgery, whereas patients with advanced-stage disease will receive neoadjuvant treatment followed by surgery.
* Ability to attend scheduled follow-up visits, if applicable, for additional peripheral blood sample collection during treatment.

Exclusion Criteria:

* Presence of any active infection or underlying condition that could compromise the safety of tissue and blood sampling.
* Prior history of another malignancy that might interfere with data interpretation related to non-small cell lung cancer progression and immune response.
* Any current use of immunosuppressive medications (e.g., high-dose steroids) which might alter immune response assessments, except as part of non-small cell lung cancer treatment.
* Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients diagnosed with non-small cell lung cancer. Individuals of diverse gender, age, and ethnicity will be included, specifically those with stage I-II and III non-small cell lung cancer, including cases with lymph node involvement.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Frequency and cytotoxic activity of patient-specific tumor-reactive T cells. | 1-30 months
  The outcome will be evaluated by measuring the percentage of tumor-reactive T cells expressing activation markers (e.g., CD137, CD107a) via flow cytometry. Cytotoxic activity will be assessed through a tumor-killing assay, quantified as the percentage of tumor cell death measured by microscopy and flow cytometry.

SECONDARY OUTCOMES:
Expression of activation, differentiation, and exhaustion markers in generated T cell product. | 12-30 months
  The outcome will be evaluated by measuring the percentage of T cells expressing activation (e.g., CD137, CD107a), differentiation (e.g., CD45RA, CCR7), and exhaustion (e.g., PD-1, TIM-3) markers via flow cytometry.

OTHER OUTCOMES:
Time required for T cell generation and functional assessment. | 18-30 months
  The outcome will be evaluated by measuring the time (in days) required to generate tumor-reactive T cells and assessing their functionality through activation marker expression (e.g., CD137, CD107a) and cytotoxic activity via flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara M Cattaneo, PhD, Principal Investigator — IRCCS Ospedale San Raffaele

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meric-Bernstam F, Larkin J, Tabernero J, Bonini C. Enhancing anti-tumour efficacy with immunotherapy combinations. Lancet. 2021 Mar 13;397(10278):1010-1022. doi: 10.1016/S0140-6736(20)32598-8. Epub 2020 Dec 4. PMID 33285141
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Rutkowski P, Lao CD, Cowey CL, Schadendorf D, Wagstaff J, Dummer R, Ferrucci PF, Smylie M, Hogg D, Hill A, Marquez-Rodas I, Haanen J, Guidoboni M, Maio M, Schoffski P, Carlino MS, Lebbe C, McArthur G, Ascierto PA, Daniels GA, Long GV, Bastholt L, Rizzo JI, Balogh A, Moshyk A, Hodi FS, Wolchok JD. Five-Year Survival with Combined Nivolumab and Ipilimumab in Advanced Melanoma. N Engl J Med. 2019 Oct 17;381(16):1535-1546. doi: 10.1056/NEJMoa1910836. Epub 2019 Sep 28. PMID 31562797
- [Background] Rosenberg SA, Restifo NP. Adoptive cell transfer as personalized immunotherapy for human cancer. Science. 2015 Apr 3;348(6230):62-8. doi: 10.1126/science.aaa4967. PMID 25838374
- [Background] Dijkstra KK, Cattaneo CM, Weeber F, Chalabi M, van de Haar J, Fanchi LF, Slagter M, van der Velden DL, Kaing S, Kelderman S, van Rooij N, van Leerdam ME, Depla A, Smit EF, Hartemink KJ, de Groot R, Wolkers MC, Sachs N, Snaebjornsson P, Monkhorst K, Haanen J, Clevers H, Schumacher TN, Voest EE. Generation of Tumor-Reactive T Cells by Co-culture of Peripheral Blood Lymphocytes and Tumor Organoids. Cell. 2018 Sep 6;174(6):1586-1598.e12. doi: 10.1016/j.cell.2018.07.009. Epub 2018 Aug 9. PMID 30100188
- [Background] Cattaneo CM, Dijkstra KK, Fanchi LF, Kelderman S, Kaing S, van Rooij N, van den Brink S, Schumacher TN, Voest EE. Tumor organoid-T-cell coculture systems. Nat Protoc. 2020 Jan;15(1):15-39. doi: 10.1038/s41596-019-0232-9. Epub 2019 Dec 18. PMID 31853056
- [Background] Cattaneo CM, Battaglia T, Urbanus J, Moravec Z, Voogd R, de Groot R, Hartemink KJ, Haanen JBAG, Voest EE, Schumacher TN, Scheper W. Identification of patient-specific CD4+ and CD8+ T cell neoantigens through HLA-unbiased genetic screens. Nat Biotechnol. 2023 Jun;41(6):783-787. doi: 10.1038/s41587-022-01547-0. Epub 2023 Jan 2. PMID 36593398
- [Background] Cattaneo CM. Identification of personalized cancer neoantigens with HANSolo. Nat Rev Cancer. 2023 Dec;23(12):800. doi: 10.1038/s41568-023-00624-z. No abstract available. PMID 37704741